CLINICAL TRIAL: NCT02999828
Title: The Safety, Immune Persistence and Consistency of Inactivated Enterovirus 71 Vaccine (Human Diploid Cell, KMB-17)
Brief Title: The Phase IVa of Inactivated Enterovirus 71 Vaccine (Human Diploid Cell, KMB-17)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Chaoyang District Centre for Disease Control and Prevention (Other); Neimenggu Province Centre for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Qihan Li, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CY2016KMEV
Record Dates: First submitted 2016-09-16; First posted 2016-12-21 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Safety of Inactivated EV71 Vaccine; Immunization of Inactivated EV71 Vaccine
Keywords: safety; immune persistence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3.0 EU in Children (Experimental): healthy children (6-71 months old) have been injected by inactivated EV71 vaccine (KMB-17) of 3.0 EU (neutralization antibodies titer unit; 100 U in phase III clinical trials, or 320 EU (Elisa assay unit) in phase I and II clinical trials)
  Interventions: Biological: inactivated EV71 vaccine (KMB-17)

INTERVENTIONS:
Biological: inactivated EV71 vaccine (KMB-17) — 3.0EU of inactivated enterovirus 71 vaccine (KMB-17) on day 0, 28.

SUMMARY:
Enterovirus 71 (EV71), a major pathogen causing hand-foot-and-mouth disease (HFMD) worldwide, is a member of the Human Enterovirus species A, family Picornaviridae. Its infection occasionally leads to severe diseases and death, with central nervous system (CNS) damage.

Recently, except of inactivated vaccine, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, such as attenuated vaccine, subunit vaccine.

A formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been finished phase I, II and III clinical trials and licensed by SFDA in China at Dec. 3, 2015. Based on the results of clinical trials, the protective efficacy of inactivated EV71 vaccine is 97% against HFMD caused by EV71. The phase IV clinical trial has been carried out from July 2016. The purpose of phase IV is to evaluated the safety and efficacy of the inactive EV71 vaccine in large scale population of Chinese children (from 6 to 71 months old).

DETAILED DESCRIPTION:
Enterovirus 71 (EV71), a major pathogen causing hand-foot-and-mouth disease (HFMD) worldwide, is a member of the Human Enterovirus species A, family Picornaviridae. Its infection occasionally leads to severe diseases and death, with central nervous system (CNS) damage.

Recently, except of inactivated vaccine, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, such as attenuated vaccine, subunit vaccine.

A formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been finished phase I, II and III clinical trials and licensed by SFDA in China at Dec. 3, 2015. Based on the results of clinical trials, the protective efficacy of inactivated EV71 vaccine is 97% against HFMD caused by EV71. The phase IV clinical trial has been carried out from July 2016. The purpose of phase IV is to evaluated the safety and efficacy of the inactive EV71 vaccine in large scale population of Chinese children (from 6 to 71 months old).

There are three parts of phase IV clinical trials have been performed. First, to evaluate the safety of the inactive EV71 vaccine in large scale population of Chinese children (from 6 to 71 months old).

Second, to evaluate the immune persistence of the inactive EV71 vaccine in large scale population of Chinese children (from 6 to 71 months old).

Third, to evaluate the efficacy of the inactive EV71 vaccine in large scale population of Chinese children (from 6 to 71 months old).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (6-71 months old children) as established by medical history and clinical examination
* The subjects' legal guardian must be aware of this vaccines
* The subjects' legal guardian voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0 ℃
* The subjects' legal guardian with the ability and objective to comply with the requirements of the protocol
* Persist for a 24-month visit (and receive blood, stool (or specimens by means of a swab) tests according to program requirements in immunogenicity observation group)
* report the HFMD cases

Exclusion Criteria:

* Subject who has a clinical diagnosis history of Hand, Foot and Mouth Disease (HFMD)
* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Severe malnutrition or dysgenopathy
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 15 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Fever before vaccination, axillary temperature ﹥37.0 ℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140 mmHg and/or diastolic blood pressure ﹥90mmHg; systolic blood pressure ﹤90 mmHg and/or diastolic blood pressure ﹤60 mmHg
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives
* take part into other vaccine or drug clinical trials in last half year

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20770 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment adverse events | Up to 24 months after finishing 2 doses immunization
  The adverse events were observed and recorded within 30 minutes post immunization (p.i.), within 0-7 days post immunization (d.p.i.) and within 8-28 d.p.i after the 1st injection, as well as after the 2nd injection. And the adverse events were also observed and recorded following within 24 months after finishing 2 doses immunization.

SECONDARY OUTCOMES:
The incidence rates of HFMD | Up to 24 months after finishing 2 doses immunization
  All hand, foot and mouth disease (HFMD) cases from the subjects were observed and recorded, including common cases, severe cases, dead cases, the cases caused by enterovirus 71, the severe cases caused by enterovirus 71, the dead cases caused by enterovirus 71. The incidence rates of the subjects from this clinical trial were calculated.
immune response of inactivated EV71 vaccine (KMB-17) in a large crowd | Up to 24 months after finishing 2 doses immunization
  The blood specimens were obtained at 0, 28, 56, 180, 360 and 720 days post the 1st immunization (p.i.). The levels of neutralization antibodies and cytokines were tested at each time point. The seroconversion rate of anti-EV71 antibodies was evaluated in serum of children. And the specific IFN-γ in subjects were tested and evaluated at 0, 180 and 360 d.p.i..

OTHER OUTCOMES:
The level of anti-EV71 antibodies was evaluated in serum of children | Up to 24 months after finishing 2 doses immunization
  The blood specimens were obtained at 0, 28, 56, 180, 360 and 720 days post the 1st immunization (p.i.). The levels of neutralization antibodies were tested at each time point. The level of anti-EV71 antibodies was evaluated in serum of children.

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, M.S., Principal Investigator — Chaoyang Provincial Center for Diseases Control and Prevention in Beijing; Shaohong Yan, M.S., Study Chair — Neimenggu Provincial Center for Diseases Control and Prevention
Locations (1):
- Chaoyang of Provincial Center for Diseases Control and Prevention in Beijing, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Participants do not agree to share individual data.